CLINICAL TRIAL: NCT04597723
Title: The Effect of Oxygen Given to Patients Undergoing Laparoscopic Cholecystectomy in the Postoperative Period on Nausea and Vomiting
Brief Title: The Effect of Oxygen Given to Patients in the Postoperative Period on Nausea and Vomiting
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Selcuk University (Other)
Collaborators: The Scientific and Technological Research Council of Turkey (Other)
Responsible Party: Principal Investigator, Tunc Tuna Pinar, PhD, Principal Investigator, Selcuk University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: Selcuk University Konya
Record Dates: First submitted 2020-10-15; First posted 2020-10-22 (Actual); Last update posted 2020-10-22 (Actual); Status verified 2020-10

CONDITIONS: Oxygen; Postoperative Nausea and Vomiting
Keywords: postoperative nausea and vomiting; Oxygen
MeSH Terms: conditions — Postoperative Nausea and Vomiting | interventions — Oxygen

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- 80% oxygen (Experimental): 80% oxygen given group
  Interventions: Drug: oxygen
- 60% oxygen (Experimental): 60% oxygen given group
  Interventions: Drug: oxygen
- routine hospital care (No Intervention): The patients in this group received routine hospital care.

INTERVENTIONS:
Drug: oxygen — Patients will be given different concentrations of oxygen.
  Arms: 60% oxygen; 80% oxygen

SUMMARY:
Carbon dioxide which is insufflated to inflate the abdominal area is absorbed from the peritoneal area and it increases endogenous catecholamines, which may consequently increase nausea and vomiting. In the literature, it is indicated that oxygen application which is one of the applications aiming to prevent nausea and vomiting is a cheap method with fewer side effects in the prevention of postoperative nausea and vomiting.

In the literature, studies on the prevention of nausea and vomiting by oxygen application in different surgical interventions have not arrived at a consensus regarding surgery type and oxygen amounts. There are studies evaluating 80% and 30% oxygen amounts in removing postoperative nausea and vomiting. Taking these conditions into consideration; the study has been planned for the purpose of examining the impact of giving 80% and 60% oxygen to patients to whom laparoscopic cholecystectomy is applied on postoperative nausea and vomiting in the postoperative period.

The study has been planned as a randomized controlled study for the purpose of determining the impact of giving oxygen (80% to the group A, 60% to the group B and control group C) to patients who apply to the general surgery service to undergo a laparoscopic cholecystectomy on postoperative nausea and vomiting in the postoperative period. The patients in the study will have the same standard anesthesia protocol and hospital routine. The study will be terminated once a total of 111 patients have been reached. In the study randomization, the patients will be assigned to the sample group according to weeks as they may influence each other. Data will be collected using Patient Introductory Information Form, which evaluates patients' socio-demographic characteristics, as well as Perioperative Period Patient Follow-Up Form and Postoperative Period Nausea-Vomiting Frequency and Severity Evaluation Form. Statistical analysis of the data to be acquired as a result of the study will be performed in the computer environment. The results to be obtained will be evaluated at p<0,05 significance level.

It is expected that the study results will provide an alternative method, which will be used in preventing the possible side effects of postoperative nausea and vomiting in patients who undergo a laparoscopic cholecystectomy. Thus, the study results may make scientific and socio-economic contributions.

DETAILED DESCRIPTION:
Postoperative nausea and vomiting; defined as any nausea, retching or vomiting. Many studies are carried out to prevent postoperative nausea and vomiting, which may be a major concern in patients undergoing surgery. However, this remains the most undesirable complication of the surgical procedure. While the incidence of postoperative nausea and vomiting is around 30% in patients receiving general anesthesia, it can rise up to 70-80% in high risk patients. Postoperative factors affecting nausea and vomiting; are grouped as factors associated with the patient, surgery, and anesthesia. Factors related to the patient; age, gender, body mass index, pain, anxiety, presence of a history of road traffic or previous postoperative nausea and vomiting history. Surgery related factors; surgery duration and type of surgery. Factors associated with anesthesia are; type and amount of anesthetic substance, ventilation type, oral intake time, and the amount of opioid taken in the postoperative period. With postoperative nausea and vomiting; Complications such as fluid-electrolyte imbalance, wound dehiscence, hemorrhage, aspiration pneumonia, delayed discharge and increased re-hospitalization rates are seen. All these complications not only increase the length of hospital stay and cost of patients, but also negatively affect the postoperative recovery quality of the patients. In addition, postoperative nausea and vomiting is an exhausting process that requires effort for caregivers. Therefore, postoperative nausea and vomiting should be prevented. Some antiemetic drugs are used to prevent nausea and vomiting, which are undesirable complications. The use of these drugs significantly increases the patient's care costs. Unlike drugs in the prevention of postoperative nausea and vomiting in the literature; It has been observed that reducing abdominal insufflation pressure, reducing anxiety in the preoperative period, acupuncture, ginger root application, alcohol sniffing, listening to music and extra oxygen therapy practices. Oxygen administration, which is one of the applications to prevent nausea and vomiting, is stated as an inexpensive method with low side effects in preventing postoperative nausea and vomiting. One of these methods is an irreversible mask. 60% with 6lt / min oxygen application with non-recyclable mask; 80% oxygen can be given from 8 lt / min. There are studies In the literature regarding the prevention of nausea and vomiting by oxygen administration. in a study they conducted on patients who underwent colon resection; They found that administration of 80% oxygen during anesthesia and for two hours after anesthesia reduced the postoperative nausea and vomiting rate from 30% to 17%. In the study conducted on gynecological patients who underwent laparoscopy, it was found that the rates of nausea and vomiting in patients who were given 80% oxygen were statistically significantly lower than those who were given 30% oxygen. Found that the rate of nausea and vomiting decreased from 28.3% to 24.5% in the group where they gave oxygen at 8 lt / min with a simple face mask for 6 hours in the postoperative period after cesarean delivery, but it was not statistically significant. . Laparoscopic cholecystectomy is the removal of the gallbladder from three or four small holes in cases where polyps and stones are problematic in the gallbladder. One of the symptoms that patients frequently complain after laparoscopic cholecystectomy is nausea and vomiting. In laparoscopic interventions applied in abdominal surgeries, the abdominal area is inflated so that the surgery can be performed comfortably, thus increasing abdominal pressure. The diaphragm is pushed up due to the increase in abdominal pressure. This situation causes the diaphragm to be more irritated. In addition, carbon dioxide insufflated to inflate the abdominal area is absorbed from the peritoneal area and increases endogenous catecholamines. In this case, nausea and vomiting may increase.

Postoperative nausea and vomiting, which prolongs the postoperative recovery period, are often seen in patients within the first 24 hours. Therefore, minimizing nausea and vomiting after laparoscopic cholecystectomy is important for the patient. In the literature, no study on oxygen administration has been found in studies conducted to relieve nausea and vomiting after laparoscopic cholecystectomy. In the studies conducted in the literature regarding the prevention of nausea and vomiting by oxygen administration in different surgical procedures, a consensus could not be reached on the type of surgery and the amount of oxygen. In addition, there are studies evaluating 80% and 30% oxygen content in relieving postoperative nausea and vomiting.Considering these situations, this research; It was planned to examine the effects of 80%, 60% and air oxygen on postoperative nausea and vomiting in patients who underwent laparoscopic cholecystectomy.

ELIGIBILITY:
Inclusion criteria

* Surgery time is 2 hours or less
* The patient does not have peripheral vascular disease
* The patient does not have a psychiatric disorder
* The patient can communicate verbally
* The patient is not using anticoagulant drugs
* The patient's hemoglobin level in the preoperative period is in the range of 12-16 g / dL
* The patient's American Society of Anesthesiologist (ASA) value is between 1-2
* The patient is not smoking
* The patient is between 18 and 65 years old
* In the intraoperative period, the carbon dioxide gas pressure used to inflate the abdomen is between 10-12.
* The patient's willingness to participate in the research
* The patient does not have respiratory diseases (such as bronchitis)
* The patient does not have claustrophobia

Exclusion Criteria

- The patient is using anticoagulant medication

Ages: 18 Years to 65 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 111 (Estimated)
Dates: Start 2022-05-03 (Estimated); Primary Completion 2023-01-03 (Estimated); Study Completion 2023-05-03 (Estimated)

PRIMARY OUTCOMES:
severity of nausea | 0-24 hours in the postoperative period
  severity of nausea was measured using a 10-cm visual analog scale, The patients were explained that 1 point indicated "no nausea" and 10 points indicated "severe nausea," and then they were asked to give 1-10 points for their severity of nausea.
severity of vomiting | 0-24 hours in the postoperative period
  severity of vomiting was measured using a 10-cm visual analog scale, The patients were explained that 1 point indicated "no vomiting" and 10 points indicated "severe vomiting," and then they were asked to give 1-10 points for their severity of vomiting

CONTACTS AND LOCATIONS:
Overall Officials: Hulya Bulut, Study Chair — Gazi University; Sevil Guler Demir, Study Chair — Gazi University; Faruk Cicekci, Study Chair — Selcuk University; Hulagu Barıskaner, Study Chair — Selcuk University; Mustafa Sahin, Study Chair — Selcuk University; Inci Kara, Study Chair — Selcuk University
Locations (1):
- Pınar tunç tuna, Konya, Turkey (Türkiye)